CLINICAL TRIAL: NCT04700904
Title: The Reliability and Validity of the PortionSize and MyFitnessPal Apps (Study 1: Laboratory-based Evaluation)
Brief Title: PortionSize Study 1 Laboratory-based Evaluation)
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, PBRC Professor, Director - Ingestive Behavior Laboratory, Pennington Biomedical Research Center
Other Study IDs: PBRC 2019-062
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to test the accuracy and user satisfaction of the PortionSize™ app and the MyFitnessPal© app during laboratory controlled test meals.

DETAILED DESCRIPTION:
Accurately quantifying food intake is vital to promoting health and reducing chronic disease risk. Food intake encompasses energy intake, nutrient intake (macronutrients, micronutrients, vitamins, minerals), and intake of various food groups (e.g., fruits, vegetables), and thus reflects the nutritional status of individuals. Nutrition affects disease risk, including risk of developing obesity, diabetes, and cancer, all of which negatively affect the United States (U.S). Nonetheless, accurate assessment of food and nutrient intake has remained challenging, despite an improvement in methods. Self report methods, namely food records, are a mainstay of nutritional epidemiology research, with food recall being another popular method. These methods rely on the participant to accurately estimate portion size and, for food recall, remember what was consumed. The accuracy of these methods have been questioned and the problems with human recall have been comprehensively outlined. As a result, there remains a significant need for methods that are sufficiently accurate to provide researchers with good outcome data and to guide health promotion efforts.

The PortionSize™ app was designed by our laboratory to overcome the limitations outlined above, and to guide users to follow specific diets. PortionSize relies on users capturing images of their food selection and waste. Food intake data are immediately provided since the user relies on built in tools, including templates, to estimate portion size. However, despite promising early indications, the PortionSize app's validity has yet to be extensively tested. Determining the accuracy of PortionSize is vital before users can utilize the app to obtain immediate feedback about their food intake. We accordingly aim to test the validity of PortionSize in a controlled laboratory setting. We will also test the validity of the MyFitnessPal© app, which is similar to an electronic food record.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-70 years
* Body mass index (BMI) 18.5 - 50
* Ownership of an iPhone model 6s or later, which the participant is willing to use for the study
* Access to Apple ID, password, and email address and willing to use them in the course of the study
* Willing to use data and any accompanying charges as part of study participation
* Willing to be re-contacted for future research and/or follow-up

Exclusion Criteria:

* Center employee
* Any condition or circumstance that could impede study completion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants ages 18 to 70 in the Baton Rouge, LA area.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center; Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lozano CP, Neubig KE, Saha S, Broyles ST, Apolzan JW, Martin CK. Validity of the PortionSize application compared with that of MyFitnessPal for accurately estimating intake: a randomized crossover laboratory-based evaluation. Am J Clin Nutr. 2024 Aug;120(2):419-430. doi: 10.1016/j.ajcnut.2024.05.023. Epub 2024 May 31. PMID 38825184

RESULTS

PARTICIPANT FLOW:
Groups:
- MyFitnessPal (V1) PortionSize (V2): MyFitnessPal app: Dietary tracking completed using a commercial-based dietary assessment application with associated website
  Portion Size app: Dietary tracking completed using a novel mobile app that relies on food photography to provide immediate feedback to the user on energy (kcals), food groups, alcohol, saturated fat, and added sugar intake.
- PortionSize (V1) MyFitnessPal (V2): Portion Size app: Dietary tracking completed using a novel mobile app that relies on food photography to provide immediate feedback to the user on energy (kcals), food groups, alcohol, saturated fat, and added sugar intake.
  MyFitnessPal app: Dietary tracking completed using a commercial-based dietary assessment application with associated website
Period: Overall Study
Arm/Group | MyFitnessPal (V1) PortionSize (V2) | PortionSize (V1) MyFitnessPal (V2)
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: all 42 participants who completed the study
Groups:
- All Participants: all 42 participants that completed the study
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Weight [Mean (Standard Deviation); unit: kg] | 81.5 (22.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Simulated Energy (kcal) Intake Between the Criterion Measure (Weighed Food) and Two Smartphone Apps (PortionSize and MyFitness Pal).
Description: The outcome variable was the difference between the criterion measure (directly weighed foods from a simulated lunch meal) and two apps: PortionSize and MyFitnessPal. The outcome measure for the PortionSize app was calculated as: energy intake values from PortionSize minus energy intake values from weighed foods. The outcome measure for the MyFitnessPal app was calculated as: energy intake values from MyFitnessPal minus energy intake values from weighed foods.
Time Frame: 2.5 hours
Population: All participants completed the study protocols using the PortionSize app and the MyFitnessPal app across two study visits (1 app at each visit). Groups defined in the participant progression section distinguish participants who used the PortionSize app first from those who used the MyFitnessPal app first.
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- PortionSize App: Dietary tracking completed using a novel mobile app that relies on food photography to provide immediate feedback to the user on energy (kcals), food groups, alcohol, saturated fat, and added sugar intake.
- MyFitnessPal App: Dietary tracking completed using a commercial-based dietary assessment application with associated website
Arm/Group | PortionSize App | MyFitnessPal App
Number analyzed (Participants) | 42 | 42
kcal | -150.1 (489.5) | 79.8 (583.3)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT04700904/Prot_SAP_000.pdf